CLINICAL TRIAL: NCT00706784
Title: Inducing a Medical Castration With a GnRH Agonist While Simultaneously Replacing Physiologic Levels and Patterns of Human Sex Steroid Hormones Using an Ethylvinyl Acetate (EVA) Vaginal Ring Delivery System
Brief Title: Ethylvinyl Acetate (EVA) Vaginal Ring Delivery System Study
Acronym: VaginalRing
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor making changes to manufacturing of vaginal ring.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Combinent (Unknown)
Responsible Party: Principal Investigator, Alexandra Kimball, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-P-001343
Record Dates: First submitted 2008-06-25; First posted 2008-06-30 (Estimated); Results first posted 2014-06-13 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
Keywords: Healthy women 18-40 years of age
MeSH Terms: interventions — Extravehicular Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Drug: Ethylvinyl Acetate (EVA) Vaginal Ring Delivery System

INTERVENTIONS:
Drug: Ethylvinyl Acetate (EVA) Vaginal Ring Delivery System — Ethylvinyl Acetate (EVA) Vaginal Ring Delivery System

SUMMARY:
This research study is looking at how well a new drug delivery system, called the vaginal ring, works to get hormones into your body as a form of birth control.

DETAILED DESCRIPTION:
3-Day Study (outpatient)

Healthy normal volunteers will participate in a 3-day outpatient study that will begin between days 1-7 of their menstrual cycle (i.e. early follicular phase). A negative urinary hCG will be obtained in these women prior to their starting the 3-day study. On the first day, subjects will have 4 baseline blood samples of 5mL each drawn at 20-minute intervals over an hour (Time = 0, +20, +40, +60). These will be pooled and will represent the pretreatment determination of gonadotropins and sex steroid levels. Thereafter, the individual vaginal rings to be tested will be inserted. Over the ensuing 3 days, subjects will have 3 blood draws per day (at approximately 8-9 AM, 12-1PM, and 4-5PM).

Serum levels of LH, FSH, E2, and P will be determined at the above time points for the next 3 days. A repeat CBC and LFT's will be done with the final blood draw. The only exceptions to this protocol will be those patients with the Sex Steroid Only rings in whom 75 ug/kg of a GnRH antagonist (Acyline IND# 58,448) will be administered subcutaneously every other day and upon subsequent onset of menses, subjects will return during day 3-6 for repeat LFT's and gonadotropins. This will ensure the return of normal liver function and hormonal levels.

A visual vaginal examination and colposcopy will be done at baseline and at the time of the removal of the ring. If lesions or abrasions are found at study termination, subjects will be followed until the lesions resolve. For the initial 3-day studies, daily visual inspection of the vaginal tissues will be conducted and findings recorded in a standardized manner.

The schedule of more intensive early sampling is selected to be certain that no rapid release of medication occurs from the rings during the earliest phase following their insertion. This will also document that we have, in fact, achieved a steady state of release of the ring's content in the circulation prior to expanding the duration of these studies to 14 days in the second portion of part A.

14 Day Study (14-Day Outpatient + 36-hour Inpatient)

Healthy normal volunteers will participate in a 14-day study that will begin between days 1-7 of their menstrual cycle (i.e. early follicular phase). A negative urinary hCG will be obtained in these women prior to their starting the 14-day study. On the first day, subjects will have 4 baseline blood samples of 5mL each drawn at 20-minute intervals over an hour (Time = 0, +20, +40, +60). These will be pooled and will represent the pretreatment determination of gonadotropins and sex steroid levels.

The individual vaginal rings to be tested will then be inserted. Subjects will return each day for the next 13 days between 8am and 12pm to the General Clinical Research Center to have 5mL of blood drawn to measure serum levels of LH, FSH, E2, and P. On day 14, the vaginal ring will be removed.

A visual vaginal examination and colposcopy will be done at baseline and at the time of the removal of the ring. If lesions or abrasions are found at study termination, subjects will be followed until the lesions resolve. For the initial 14-day studies, visual inspection of the vaginal tissues will be conducted at least 3 times per week and findings recorded in a standardized manner.

Two days later, subjects will be admitted to the General Clinical Research Center between the hours of 8am and 12pm for a 36-hour inpatient stay. Subjects will be given a 240 ug dose of the GnRH agonist intravenously and the subject's bloods drawn for GnRHa determinations at 0, 15, 30, 60, 75, 90, 120min, and then hourly for the remaining 36 hours. A repeat cbc will be drawn with the final blood draw.

These determinations will then be compared to the GnRH agonist determinations from the vaginal route of delivery during the previous 14 days and hence the % absorption of the GnRHa from the vagina.

The exceptions to this protocol will be those patients with the Sex Steroid Only rings in whom 75 ug/kg of a GnRH antagonist (Acyline IND# 58,448) will be administered subcutaneously every other day for the course of the 14 days. These subjects will not undergo the inpatient stay after the ring is removed. Repeat LFT's will be drawn with the final blood draw as well. Anytime the Acyline injection is given, subjects will be monitored for at least 30 minutes after each injection for signs/symptoms of an allergic reaction. Upon subsequent onset of menses, subjects will return during days 3-6 for repeat LFT's and gonadotropins. This will ensure the return of normal liver function and hormonal levels.

ELIGIBILITY:
Inclusion Criteria:

1. A history of normal regular menstrual cycles (25-35 days);
2. A normal physical examination;
3. A body mass index (BMI) between 19 & 29
4. A normal CBC, normal Prolactin level, normal LFT's
5. A negative urinary hCG at the initiation of each study; and
6. An agreement to refrain from attempting to conceive during the experimental cycle and the cycle thereafter by either abstinence and/or use of a barrier method of contraception.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2008-06; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra B. Kimball, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Clinical Unit for Research Trials In Skin (CURTIS), Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 18 mg Leuprolide for 3 Days | 36 mg Leuprolide for 3 Days
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 18 mg Leuprolide for 3 Days | 36 mg Leuprolide for 3 Days | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Serum Leuprolide Levels After EVA Ring Transvaginal Drug Delivery System Insertion
Time Frame: 8 hours
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | 18 mg Leuprolide for 3 Days | 36 mg Leuprolide for 3 Days
Number analyzed (Participants) | 3 | 3
pg/ml | 310 (221) | 1220 (735)

ADVERSE EVENTS:
Time Frame: 3 days
Arm/Group | 18 mg Leuprolide for 3 Days | 36 mg Leuprolide for 3 Days
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 2/3 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 18 mg Leuprolide for 3 Days (N=3) | 36 mg Leuprolide for 3 Days (N=3)
Displacement of Vaginal Ring (Reproductive system and breast disorders) | 2 (2) | 0 (0) — Two subjects reported displacement of the vaginal ring associated with Valsava (forceful exhalation with a closed nose and mouth).

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No